CLINICAL TRIAL: NCT06680271
Title: Exercise Prescription Via Telerehabilitation for Older Adults With Cardiopulmonary Disease in Antioquia, Colombia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Universitaria Maria Cano (Other)
Responsible Party: Principal Investigator, Silvia Patricia Betancur Bedoya, Professor, Universidad Iberoamericana A.C., Mexico
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-222
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Telerehabilitation; Exercise; Noncommunicable Disease
Keywords: Telerehabilitation; Physical Activity
MeSH Terms: conditions — Motor Activity; Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: The intervention group will consist of 25 subjects receiving a multicomponent physical exercise intervention (aerobic, strength, flexibility, and neuromotor) delivered by a physical therapist via the Microsoft Teams platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth interventions (Experimental): The intervention group will consist of 25 subjects receiving a multicomponent physical exercise intervention (aerobic, strength, flexibility, and neuromotor) delivered by a physical therapist via the Microsoft Teams platform.
  Interventions: Other: Remote exercise
- Home Intervention (Active Comparator): The control group will consist of 25 subjects receiving traditional physical therapy at home from a physical therapist
  Interventions: Other: Home exercise

INTERVENTIONS:
Other: Remote exercise — The intervention group will consist of 25 subjects receiving a multicomponent physical exercise intervention (aerobic, strength, flexibility, and neuromotor) delivered by a physical therapist via the Microsoft Teams platform
  Arms: Telehealth interventions
Other: Home exercise — The control group will consist of 25 subjects receiving traditional physical therapy at home from a physical therapist.
  Arms: Home Intervention

SUMMARY:
Objective: To evaluate the effects of telerehabilitation with physical exercise in older adults with cardiorespiratory disease in Antioquia, Colombia.

Methods: This study will be a single controlled trial conducted at a single center. A sample of 50 older adults with cardiorespiratory diseases will be included. The intervention group will consist of 25 subjects receiving a multicomponent physical exercise intervention (aerobic, strength, flexibility, and neuromotor) delivered by a physical therapist via the Microsoft Teams platform. The control group will consist of 25 subjects receiving traditional physical therapy at home from a physical therapist. The intervention will be pre-registered on "ClinicalTrials.gov".

Expected Results: An improvement in quality of life, measured by the WHOQOL-Bref (World Health Organization Quality of Life), an increase in physical condition assessed with the Senior Fitness Test battery, and a reduction in frailty measured by the Short Physical Performance Battery (SPPB) are expected. Additionally, the development of a cardiopulmonary telerehabilitation protocol is anticipated.

DETAILED DESCRIPTION:
This study will explore the effects of prescribing physical exercise through telerehabilitation for older adults with cardiorespiratory diseases in Antioquia, Colombia. It will aim to determine which exercise prescriptions are most beneficial and feasible for this population within a telerehabilitation model, taking into account the specific conditions they face.

The study will address three main questions. First, it will identify which types of physical exercises are most suitable for older adults with various cardiorespiratory conditions when delivered via telerehabilitation. Second, it will examine how to best implement these exercises to ensure safety, engagement, and effectiveness through remote guidance. Finally, the study will evaluate the benefits of telerehabilitation-prescribed physical exercises, particularly regarding improvements in quality of life for older adults managing these health conditions.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participate in the study.
* Inclusion will be considered for individuals with specific chronic medical conditions, including Chronic Obstructive Pulmonary Disease (COPD), which will be diagnosed according to the guidelines established in the widely used Global Initiative for Chronic Obstructive Lung Disease (GOLD) guide in clinical and research contexts. Similarly, asthma will be included, identified according to the criteria outlined in the Global Initiative for Asthma (GINA) guide. Heart failure will also be included, categorized based on the New York Heart Association (NYHA) functional classification previously validated in Colombian populations. Additionally, metabolic syndrome will be included, with confirmation based on criteria defined by the World Health Organization (WHO).
* The patient's diagnosis must be confirmed through medical history.
* These specific criteria will guide the selection of participants who meet the established requirements for this study.
* Must be able to communicate verbally or in writing.
* Must be in a stable phase of their illness, supported by medical history.
* A minimum of 3 months of illness for the condition to be considered chronic.
* Patients with Type II Diabetes Mellitus must have a glucose level lower than 200 mg/dL during the tele-rehabilitation session.

Exclusion Criteria:

* Dementia.
* Epilepsy or a history of seizures.
* Patient who has recently undergone surgery.
* Delirium.
* Acute myocardial infarction or recent unstable angina.
* Uncontrolled atrial or ventricular arrhythmias.
* Dissecting aortic aneurysm.
* Severe aortic stenosis.
* Acute endocarditis/pericarditis.
* Uncontrolled hypertension.
* Acute thromboembolic disease.
* Severe acute heart failure.
* Severe acute respiratory failure.
* Uncontrolled orthostatic hypotension.
* Diabetes mellitus with acute decompensation or uncontrolled hypoglycemia.
* Recent fracture (within the last month, strength training).
* Any other circumstance deemed by the evaluator or the subject that prevents physical activity.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life - BREF (WHOQOL-BREF) | Month 1 vs Month 3
  The WHOQOL-BREF is a 26-item questionnaire covering four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items), along with items on overall quality of life and general health. Each item is rated on a 5-point ordinal scale, and scores are linearly transformed to a 0-100 scale.

SECONDARY OUTCOMES:
Frailty SPPB (Short Physical Performance Battery) | Month 1 vs Month 3
  The SPPB will assess lower limb function through five tests covering balance, strength, and mobility. Balance tests will have three progressively challenging stages (feet together, semi-tandem, and full tandem), aiming for 10 seconds unaided at each stage. Gait speed will be measured with a portable gait analysis system. For the "five times sit-to-stand" test, participants will begin seated and, after demonstrating one sit-to-stand, will complete five repetitions as quickly as possible, with feet flat on the floor. Scores will reflect performance, with a maximum score of 12; lower scores indicate greater frailty in older adults.
Senior Fitness Test- Physical Condition | Month 1 vs Month 3
  The Senior Fitness Test evaluates various physical fitness components for older adults:
  Lower Body Strength - Chair Stand Test (30 seconds): Measures leg strength by counting how many times a person can rise from a chair in 30 seconds. More repetitions are better.
  Upper Body Strength - Arm Curl Test: Counts how many arm curls can be completed in a set time (30 seconds). More repetitions are better.
  Aerobic Endurance - 6-Minute Walk Test: Assesses walking endurance over 6 minutes, measured in meters. More meters walked are better.
  Upper Body Flexibility - Back Scratch Test: Measures shoulder flexibility by attempting to touch hands behind the back. Greater reach is better.
  Lower Body Flexibility - Chair Sit and Reach Test: Assesses flexibility of the hamstrings and lower back, measured in centimeters. Greater reach is better.

CONTACTS AND LOCATIONS:
Locations (1):
- Silvia Betancur, Envigado, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in telerehabilitation
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will be made accessible for up to 24 months.
Access Criteria: Access to trial Individual Patient Data (IPD) is available to qualified researchers conducting independent scientific research. Requests will be granted after review and approval of a research proposal. For more information or to submit a request, please contact principal researcher.